CLINICAL TRIAL: NCT01038037
Title: A Phase II Study of First-Line Chemotherapy and Panitumumab in Advanced NSCLC Selected by Mutational Status
Brief Title: First-Line Chemotherapy and Panitumumab in Advanced Non-Small Cell Lung Cancer
Acronym: Lung-TRIO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 1. Very low enrollment rate.
  2. Recent studies question the effect of adding panitumumab in this category of patients.
  3. Too high toxicity rate
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2009-015068-32
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; Non small cell lung cancer; Triple mutational status; KRAS; BRAF; PI3K
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; Vinorelbine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Carboplatin — i.v. day 1: AUC 5 x (GFR + 25) mg q3w
Drug: Vinorelbine — i.v. day 1: 30 mg/m2 q3w Orally day 8: 60 mg/m2 q3w
Drug: panitumumab — i.v. day 1: 9 mg/kg q3w

SUMMARY:
The purpose of this study is to determine whether the addition of panitumumab to standard chemotherapy in first-line treatment of advanced Non Small Cell Lung Cancer improves the treatment outcome. Patients are selected based on triple mutational status.

DETAILED DESCRIPTION:
Advanced NSCLC holds a very poor prognosis with a moderate response rate to standard chemotherapy. The standard first-line treatment for advanced NSCLC is platinum based combination chemotherapy. The response rates are less than 30% and a substantial amount of patients will experience unnecessary toxicity in terms of e.g. nausea, vomiting, neuropathies or a considerable risk of renal toxicity. The median progression free survival is 3-4 months and consequently, the median overall survival is less than one year (Hotta et al 2007). Addition of new biological agents to standard chemotherapy regimens may improve the outcome for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic (stage IV) NSCLC
* Measurable disease according to RECIST v.1.0 2009
* KRAS, BRAF and PI3K wild type in primary tumor or metastatic tissue.
* Age ≥18
* PS < 2
* Adequate organ function

Haematology:

* Neutrophil count ≥1.5x10^9/L
* Platelet count ≥100x10^9/L
* Leucocyte count > 3,000/mm

Hepatic function:

* Total bilirubin ≤ 1.5 times the upper normal limit (UNL)
* Serum transaminases ≤ 2.5xUNL in absence of liver metastases, or ≤ 5xUNL in presence of liver metastases

Renal Function:

* Creatinine clearance ≥ 50 mL/min and serum creatinine ≤ 1.5xUNL

Metabolic function:

* Magnesium ≥ lower limit of normal.
* Calcium ≥ lower limit of normal.

Consent to translational research studies

Written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment/randomization, active severe infections or other concurrent disease.
* Known CNS metastasis (pretreatment routine assessment not required)
* Prior chemotherapy for metastatic disease
* Indication for radiation therapy or prior radiotherapy within 30 days before treatment start.
* Other malignant diseases within 5 years prior to inclusion in the study, except basal cell squamous carcinoma of the skin and cervical carcinoma-in-situ.
* Other experimental therapy within 30 days prior to treatment initiation.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Patients pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Patients (male or female) not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 3 years

SECONDARY OUTCOMES:
Progression free survival | Up to 3 years
Overall survival | Up to 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Vejle Hospital, Vejle, Denmark